CLINICAL TRIAL: NCT02342522
Title: Effect of Remote Ischaemic Conditioning on Clinical Outcomes in ST-segment Elevation Myocardial Infarction Patients Undergoing Primary Percutaneous Coronary Intervention (CONDI2/ERIC-PPCI)
Brief Title: Effect of Remote Ischaemic Conditioning on Clinical Outcomes in STEMI Patients Undergoing PPCI (CONDI2/ERIC-PPCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: British Heart Foundation (Other); London School of Hygiene and Tropical Medicine (Other); King's College London (Other); Oxford University Hospitals NHS Trust (Other); University of Aarhus (Other); Rigshospitalet, Denmark (Other); Aalborg University Hospital (Other); Odense University Hospital (Other); Hospital Universitario Central de Asturias (Other); Clinical Centre of Serbia (Other); Military Medical Academy, Belgrade, Serbia (Other); Central Denmark Region (Other); Region of Southern Denmark (Other); Prehospital Emergency Medical Service, The North Denmark Region (Unknown); Region Zealand (Other); The Danish Medical Research Council (Other); Aarhus University Hospital (Other); North Cumbria University Hospitals NHS Trust (Other); Barts & The London NHS Trust (Other); Mid and South Essex NHS Foundation Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); Manchester University NHS Foundation Trust (Other Government); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); The Royal Wolverhampton Hospitals NHS Trust (Other Government); Royal Free Hospital NHS Foundation Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); East and North Hertfordshire NHS Trust (Other Government); Portsmouth Hospitals NHS Trust (Other Government); United Lincolnshire Hospitals NHS Trust (Other); Papworth Hospital NHS Foundation Trust (Other Government); Blackpool Victoria Hospital (Other); Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (Other Government); Brighton and Sussex University Hospitals NHS Trust (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); University Hospitals of North Midlands NHS Trust (Other); Heart of England NHS Trust (Other); Kettering General Hospital NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); East Kent Hospitals University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS/14/3/31002; NCT01857414 (obsolete NCT alias)
Record Dates: First submitted 2014-10-20; First posted 2015-01-21 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2018-10

CONDITIONS: STEMI; Myocardial Reperfusion Injury
Keywords: Cardioprotection; STEMI; PPCI; Myocardial reperfusion injury; Myocardial infarct size; ST-elevation myocardial infarction; Remote Ischaemic Conditioning; Cardiovascular mortality
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote ischemic conditioning (Active Comparator): AutoRIC device will be placed on the upper arm and an active RIC protocol will be delivered (4x5 min cycles of inflation to 200mmHg and deflation) prior to PPCI.
  Interventions: Device: Remote ischemic conditioning
- Sham control (Sham Comparator): Sham AutoRIC device will be placed on the upper arm and a sham RIC protocol will be delivered prior to PPCI.
  Interventions: Device: Control

INTERVENTIONS:
Device: Remote ischemic conditioning — An automated autoRIC™ cuff will be placed on the upper arm and inflated to 200mmHg for 5 minutes and then deflated for 5 minutes, a cycle which will be undertaken 4 times in total.
  Arms: Remote ischemic conditioning
Device: Control — An automated autoRIC™ cuff will be placed on the upper arm and a simulated inflation and deflation protocol will be applied.
  Arms: Sham control

SUMMARY:
The purpose of this study is to determine whether remote ischemic conditioning can reduce cardiac death and hospitalization for heart failure at 12 months in patients presenting with a ST-elevation myocardial infarction and treated by percutaneous coronary intervention.

DETAILED DESCRIPTION:
The CONDI2/ERIC-PPCI trial is a randomised controlled clinical trial investigating whether remote ischemic conditioning (RIC) can reduce cardiac death and hospitalization for heart failure at 12 months in 5400 patients presenting with a ST-elevation myocardial infarction (STEMI) and treated by percutaneous coronary intervention (PPCI).

ELIGIBILITY:
Inclusion criteria:

1. Onset of STEMI symptoms within 12 hours, lasting for more than 30 minutes
2. Patients older than 18 years
3. Suspected STEMI (ST-elevation at the J-point in two contiguous leads with the cutoff points: ≥0.2 millivolt (mV) in men or ≥0.15 mV in women in leads V2-V3 and/or ≥0.1 mV in other leads)

Exclusion criteria:

1. Previous coronary artery bypass graft surgery
2. Myocardial infarction within the previous 30 days
3. Treatment with thrombolysis within the previous 30 days
4. Left bundle branch block
5. Patients treated with therapeutic hypothermia
6. Conditions precluding use of RIC (paresis of upper limb, use of an a-v shunt)
7. Life expectancy of less than 1 year due to non-cardiac pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5413 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Rates of cardiac death and hospitalization for heart failure (HHF) at 1 year. | One year

SECONDARY OUTCOMES:
Rates of cardiac death and HHF at 30 days. | 30 days
Rates of all-cause death, repeat coronary revascularisation, reinfarction, stroke at 30 days and 12 months. | 12 months
TIMI flow post-PPCI. | 1 week
Quality of life at 6-8 weeks and 12 months (EuroQol EQ-5D-5L). | One year
Biomarkers substudy: Enzymatic infarct size - 48 hour area-under-the-curve (AUC) cardiac biomarkers | 1 week
CMR substudy: Cardiac MRI in first week and at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Derek Hausenloy, MD PhD, Principal Investigator — The Hatter Cardiovascular Institute, University College London; Hans Erik Botker, MD PhD, Principal Investigator — University of Aarhus
Locations (35):
- Denmark (7):
  - Prehospital Emergency Medical Service, North Denmark Region, Aalborg
  - Aalborg University Hospital, Aalborg
  - Prehospital Emergency Medical Service, Central Denmark Region, Aarhus
  - Prehospital Emergency Medical Service, Region Zealand, Ballerup Municipality
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
  - Prehospital Emergency Medical Service , South Denmark Region, Vejle
- Clinical Centre of Serbia, Belgrade, Serbia
- Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias, Spain
- United Kingdom (26):
  - Royal Sussex County Hospital, Brighton, Sussex
  - William Harvey Hospital, Ashford
  - Basildon University Hospital, Basildon
  - Birmingham Heartlands Hospital, Birmingham
  - Blackpool Victoria Hospital, Blackpool
  - Royal Bournemouth Hospital, Bournemouth
  - Bristol Royal Infirmary, Bristol
  - Papworth Hospital, Cambridge
  - Cumberland Infirmary, Carlisle
  - Coventry University Hospital, Coventry
  - Kettering General Hospital, Kettering
  - Leeds General Infirmary, Leeds
  - Lincoln County Hospital, Lincoln
  - Hammersmith Hospital, London
  - Kings College London Hospital, London
  - St Bartholomew's Hospital, London
  - St Thomas Hospital, London
  - The Royal Free Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Norfolk and Norwich University Hospital, Norwich
  - John Radcliffe Hospital, Oxford
  - Queen Alexandra Hospital, Portsmouth
  - Northern General Hospital, Sheffield
  - Lister Hospital, Stevenage
  - Royal Stoke University Hospital, Stoke-on-Trent
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hausenloy DJ, Kharbanda RK, Moller UK, Ramlall M, Aaroe J, Butler R, Bulluck H, Clayton T, Dana A, Dodd M, Engstrom T, Evans R, Lassen JF, Christensen EF, Garcia-Ruiz JM, Gorog DA, Hjort J, Houghton RF, Ibanez B, Knight R, Lippert FK, Lonborg JT, Maeng M, Milasinovic D, More R, Nicholas JM, Jensen LO, Perkins A, Radovanovic N, Rakhit RD, Ravkilde J, Ryding AD, Schmidt MR, Riddervold IS, Sorensen HT, Stankovic G, Varma M, Webb I, Terkelsen CJ, Greenwood JP, Yellon DM, Botker HE; CONDI-2/ERIC-PPCI Investigators. Effect of remote ischaemic conditioning on clinical outcomes in patients with acute myocardial infarction (CONDI-2/ERIC-PPCI): a single-blind randomised controlled trial. Lancet. 2019 Oct 19;394(10207):1415-1424. doi: 10.1016/S0140-6736(19)32039-2. Epub 2019 Sep 6. PMID 31500849